CLINICAL TRIAL: NCT03842579
Title: Effects of High-protein Diet Combined With Exercise to Counteract Frailty in Pre-frail and Frail Community-dwelling Older Adults: a Three-arm Randomized Controlled Trial
Brief Title: Protein and Exercise to Counteract Frailty in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Metropolitan University College (Other); Municipality of Odense, Denmark (Unknown); Arla Foods (Industry)
Responsible Party: Principal Investigator, Paolo Caserotti, Professor and Head of Center for Active and Healthy Ageing, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20180048; S-20180048 (Other: Regional Committee Health Research Ethics, Southern Denmark)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Physical Frailty
Keywords: Frailty; Ageing; High-Protein diet; Protein Supplementation; Resistance Training; Strength Training; Muscle Power; Muscle Strength; Muscle Mass; Functional Performance; Nutritional Status
MeSH Terms: conditions — Frailty | interventions — Resistance Training; Diet, High-Protein; Health Planning Guidelines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not be informed about allocation of the participants prior to the assessment of outcomes. The participants will be informed not to give any information to outcome assessors about the result of their randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise and Protein (EXEPROT) (Experimental): Participants in EXEPROT receive: a high-protein diet combined with Resistance training. The high-protein diet is based on milk-based protein-rich products to supplement the habitual diet (corresponding to a protein intake of 1.5 g/kg/day). 4-day food records are used to estimate the needed protein. Of the shelf-products (e.g. milk, cheese) are used considering the individually preferences. Products are delivered once a week. The training intervention includes progressive explosive type heavy-resistance training two times per week. The intervention runs for 16 weeks. Adherence to the training protocol is monitored at each session. Adherence with the nutrition protocol is monitored daily plus at phone follow-ups where participants are asked about e.g. appetite, weight, habitual intake.
  Interventions: Other: Resistance training; Other: High-protein diet
- Protein-only (PROT) (Active Comparator): Participants in PROT-group receive the nutritional intervention: The high-protein diet.
  The diet is based on daily milk-based protein-rich products to supplement the habitual diet (corresponding to a total protein intake of 1.5 g/kg/day). The needed amount of protein supplementation is estimated from 4-day food records. Of the shelf-products (e.g. milk, skyr, cheeses) are used considering the individually preferences. Products will be delivered once a week at the home of the participant. The intervention runs for 16 weeks.
  Adherence with the nutrition protocol is monitored daily (registration of compliance with the dietary plan) as well as at phone follow-ups where participants are asked about e.g. changes in appetite, weight, and habitual intake.
  Interventions: Other: High-protein diet
- Recommendations (REC) (Active Comparator): Participants in the REC-Group receive the comparative intervention: Recommendations.
  The official national dietary recommendations for adults >65 years, developed by the Ministry of Environment and Food of Denmark, and related materials is given to the participants and they are encouraged to follow the guidelines (recommending a protein intake of 1.0-1.3 g/kg/day). The intervention runs for 16 weeks.
  During the intervention all groups will receive two seminars on specific topics related to healthy ageing (e.g. talks on physical activity, sedentary behaviour, and nutrition).
  Interventions: Other: Recommendations

INTERVENTIONS:
Other: Resistance training — Supervised progressive explosive type heavy-resistance training two times per week
  Arms: Exercise and Protein (EXEPROT)
Other: High-protein diet — Daily supplementation with milk-based protein-rich products
  Arms: Exercise and Protein (EXEPROT); Protein-only (PROT)
Other: Recommendations — Provided with the official national recommendations on nutrition
  Arms: Recommendations (REC)

SUMMARY:
The purpose of this study is to determine the effects of interventions with high-protein diet alone or in combination with resistance training on muscle mechanical function (muscle power and strength), frailty status, functional performance, muscle mass and quality of life.

DETAILED DESCRIPTION:
Study design: two-phase randomized controlled trial with three arms.

Phase 1 stabilization phase lasting one month. Participants with low protein intake (<1.0 g/kg/day) are provided with national guidelines for daily protein intake and publicly available information material and recommended to increase their protein intake to meet the guidelines. Compliance to the recommendation/ guidelines (eating >1.0 g/kg/day) will be evaluated by 4-day food records at the end of the stabilization phase. Only compliant participants are eligible for phase 2. Participants that are not compliant will be followed as "natural observational group" but will not be considered for the primary statistical analysis. Data collection in these participants will only include assessment of selected demographic, functional and nutritional parameters and semi-structured interviews to identify potential barriers for not improving protein intake. Semi-descriptive data will be presented if possible.

Phase 2: Three-arm randomized controlled trial lasting four months:

i) Protein-only (PROT): participants will receive milk-based protein-rich products with the aim of targeting a daily protein intake of 1.5 g/kg; ii) Exercise and Protein (EXEPROT): participants will receive the protein intervention as in the PROT-group combined with progressive explosive type heavy-resistance strength training two times per week iii) Recommendations (REC) participants receive the national nutritional recommendations for older adults and are recommended to follow these recommendations over the course of the study.

Nutritional data will be collected pre and post the stabilization phase. Collection of the primary and secondary outcomes will occur at baseline (pre phase 2) and at the 4-month follow-up (post phase 2). Nutritional assessment will also be evaluated halfway, at the 2-month follow-up.

Compliance Adherence to the exercise protocol and protein supplementation is recorded during the study. For the exercise protocol adherence will be considered as achieving minimum to 75% of valid training sessions, considered as minimum 70% of the exercises planned for each session. For the protein supplementation, adherence will be evaluated as daily protein intake of ≥ 1.35 g/kg (estimated from 24 hours recall and four-day food records) at the 2-month follow-up and at the 4-months follow-up. Compliance will also be estimated from during each delivery of products with a set of questions (e.g. how much of the supplement is consumed? Any changes to the habitual food intake?) and regular phone follow-ups. If participants are unable to reach the protein target additional face to face or phone interview will be planned to support adherence. For the REC-group adherence is defined as following the recommended intake of protein (1.0-1.3 g/kg/day).

Sample size and statistics Lower leg muscle power is the primary outcome of this study. Due to lack of studies similar to this study design (e.g. age and frailty status of the participants, type of exercise and level of protein supplementation) the investigators have calculated sample size using a combination of studies and methods. Based on findings from a 2017 study the effect of 12-weeks of protein supplementation (two daily supplements of 20 g milk protein) in combination with resistance training in +80-year-old healthy adults increased muscle power by 15% (SEM ± 5%) in comparison with -7% (SEM ± 6%) in the control group (receiving protein supplementation only). A result from a 2018 study indicate that 12 weeks of nutritional supplementation (0.8 g/kg/day, 1.2 g/kg/day or 1.5 g/kg/day) to pre-frail or frail older adults >70 years resulted in an increase in muscle mass (estimated by Dual energy X-ray Absorptiometry, DXA) of approximately 4% in the group receiving 1.5 g/kg/day. Unpublished data from the investigators research group show that change in muscle mass (estimated by DXA) accounted for 1,95% of the change in muscle power in older adults following 12 weeks of resistance training. Hence, the estimated effect of an increase in muscle mass of 4% on muscle power is 7,8%. Adding this to the results from the 2017 study gives an estimated change on 0,8% in the PROT-group. Assuming, that the change in muscle mass are comparable in the three groups the investigator therefore expect a change in muscle power of 15%, 0,8% and -7% with a standard deviation (SD) of 30 in the EXEPROT-, PROT- and REC-group, respectively.

Setting a power of 0.8 sample size with 37 participants in each arm should be enough to detect a significant difference in muscle power (significance level at 0.05). Adding 25% to account for dropouts a total of 150 participants is needed.

Intention-to-treat analysis will be performed. In addition, per-protocol analysis of participants that are compliant to the protocol will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults ≥ 80 years
* Pre-frail or frail (evaluated by the physical frailty questionnaire, SHARE-FI75+)
* Intact cognitive function (Mini Mental State Evaluation ≥4)
* Medically stable evaluated by medical screening including blood sample
* Able to participate in group-based exercise without personal assistance
* Able to understand, read and write Danish

Exclusion Criteria:

* Allergic/ intolerant to the interventions (kidney diseases, lactose intolerance etc.)
* On a weight losing diet

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline lower leg muscle power at 4 months | Baseline and 4-month follow-up
  Lower leg muscle power will be assessed unilaterally using the Nottingham Leg Rig

SECONDARY OUTCOMES:
Changes from baseline physical frailty status at 4 months | Baseline and 4 months follow-up
  Changes in frailty status will be evaluated by the physical frailty questionnaire (SHARE-FI75+) and the slightly modified version of the Frailty Phenotype assessment tool developed by Fried.
Changes from baseline countermovement jump muscle power at 4 months | Baseline and 4-month follow-up
  Weight-bearing multi-joint motor task, countermovement jump, with a linear encoder.
Changes from baseline leg press and handgrip muscle strength at 4 months | Baseline and 4-month follow-up
  Lower limb muscle strength will be measured during a maximal voluntary isometric leg press test (MVC). Subjects are seated in a custom-built unilateral leg press device (knee and ankle angles of 120 and 90, respectively) while pushing against a fixed instrumented force plate as hard and fast as possible with the dominant leg against. Muscle strength, contractile Rate of Force Development (RFD) and impulse will be determined in the trial with the highest resultant peak force.
  Handgrip: Maximal isometric handgrip strength will be assessed unilaterally using a handheld dynamometer
Changes from baseline Short Physical Performance Battery test at 4 months | Baseline and 4-month follow-up
  Physical function will be measured with the Short Physical Performance Battery (SPPB) which consists of three items (balance, 3 or 4 meters walking and repeated chair rise). Score ranges from 0-12 (each item has a score between 0 and 4).
Eating Symptom Questionnaire | Baseline
  Evaluated by a validated eating ability questionnaire. For each symptom participant range from none to severe.
Risk of Dysphagia | Baseline
  Evaluated by a validated questionnaire, the EAT-10. Resulting in a score ranging from 0-40
Appetite | Baseline
  Evaluated by a validated questionnaire the Simplified Nutritional Appetite Questionnaire. Score range from 4-20.
Changes from baseline anthropometry waist and hip circumference at 4 months | Baseline and 4 months follow-up
  Waist and hip circumference (cm) will be measured using a standard ruler.
Changes from baseline body weight at 4 months | Baseline and 4 months follow-up
  Body weight will be measured to using a transportable scale. Participants will be measured without shoes and wearing light clothing.
Changes from baseline lean and fat mass at 4 months | Baseline and 4 months follow-up
  Changes in lean mass and fat mass will be estimated by Bioelectrical Impedance Analysis.
Changes from baseline lean and fat mass and bone mineral density) to 4 months | Baseline and 4 months follow-up
  Changes in body composition (lean and fat mass and bone mineral density) will be measured by Dual-energy X-ray Absorpmetry.
Changes from baseline Health-related quality of life to 4 months | Baseline and 4-months follow-up
  Health-related quality of life questionnaires (EQ-5D-3L and SF-12) will be used. Scores range from 11111-33333 and 0-100, respectively.
Changes from baseline pain to 4 months | Baseline and 4-months follow-up
  Pain will be assessed by validated questionnaires (The brief pain inventory & Back and Neck pain survey questionnaire). Visual analogue scale (score 0-10) is combined with questions about intensity and frequency of pain.
Changes from baseline fatigue and fatigability to 4 months | Baseline and 4-months follow-up
  Validated questionnaires will be used to assess fatigue and fatigability (Mobility Fatigue, Mob-T, & The Pittsburgh Fatigability Scale). Scores ranging from 0-6 and 0-50, respectively.
Changes from baseline activities of daily living to 4 months | Baseline and 4-months follow-up
  Activities of daily living will be assessed with self-report questionnaires.
Changes from baseline fear of falling to 4 months | Baseline and 4-months follow-up
  Validated questionnaire will be used to assess fear of falling (the Falls Efficacy Scale - International). Score range from 16-64.
Changes from baseline Blood markers to 4 months | Baseline and 4-months follow-up
  Analysis of changes in markers of health and disease will be performed, e.g. Lipid profile, Hormonal profile, protein-markers of inflammation (e.g. High Sensitive C-Reaktivt Protein (HS-CRP), soluble urokinase plasminogen activating receptor (suPAR)), vitamins and minerals.
Chenages from baseline Objective measures of Physical activity, sedentary behaviour, nap and sleep to 4 months | Baseline and 4-months follow-up
  Accelerometry methodology: level and patterns of physical activity (PA), sedentary behaviour (SB), nap and sleep (NAS) will be assessed with commercially available accelerometers (e.g. Axivity, Actigraph) placed on different anatomic locations (e.g. thigh, hip) for one week.
Changes from baseline Self-reported Physical activity & sedentary behaviour to 4 months | Baseline and 4-months follow-up
  Self-report questionnaire will be used to assess physical activity and sedentary behaviour (e.g. sedentary behaviour questionnaires).
Changes from baseline Dietary intake to 4 month | Baseline and 4-months follow-up
  Dietary intake is estimated by Four-day food records and food frequency questionnaires. Protein intake is calculated as average g/day and g/kg/day.
24 hours recall | pre phase 1
  Dietary intake is estimated from 24 hours recall. Protein intake is calculated as average g/day and g/kg/day.
Changes from baseline Walking speed to 4 months | Baseline and 4 months follow-up
  Self-selected and maximal walking speed is measured.
Changes from baseline Stand and reach to 4 months | Baseline to 4 months follow-up
  The ability to stand and reach is tested
Changes from baseline Walking distance to 4 months | Baseline and 4 months follow-up
  The distance walked during 2- and 6-minutesis tested.
Changes from baseline Upper body ball throwing to 4 months | Baseline to 4 months follow-up
  The ability to throw a ball, using the upper body is tested.
Changes from baseline Rising from laying position to 4 months | Baseline to 4 months follow-up
  the ability to rise from laying position is tested.
Changes from baseline Nutritional status to 4 months | Baseline and 4 months follow-up
  Nutrititional status is estimated by validated questionnaires: the Mini Nutritional Assessment and Eating Validation Scheme. Scores range from 0-30 and 0-3, respectively.
Changes in Risk of poor protein intake to 4 months | Baseline and 4 months
  The questionnaire (protein screener) is used to estimate the probability score of having a low protein intake.

OTHER OUTCOMES:
Cognitive function | Baseline and 4-months follow-up
  The Digit Symbol Substitution Test
Gender | Baseline
  Gender (male female)
Age | Baseline
  Age (years)
Education | Baseline
  Self-report education will be assessed as number of years spent in school and maximum level of education achieved.
Marital status | Baseline
  Marital status will be evaluated as self-report.
Depression | Baseline
  depression will be evaluated with validated questionnaire at baseline (Geriatric Depression
Incontinence | Baseline
  Incontinence will be evaluated with the International Consultation on Incontinence Questionnaire (ICIQ) questionnaire at baseline (max score 21)
Chronic conditions | Baseline
  Number and type of chronic conditions will be assessed as self-report
Use of medicine | Baseline
  Direct count of name and dose of medicines performed under medical screening. The participant will be asked to bring the medicines.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caserotti, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bechshoft RL, Malmgaard-Clausen NM, Gliese B, Beyer N, Mackey AL, Andersen JL, Kjaer M, Holm L. Improved skeletal muscle mass and strength after heavy strength training in very old individuals. Exp Gerontol. 2017 Jun;92:96-105. doi: 10.1016/j.exger.2017.03.014. Epub 2017 Mar 28. PMID 28363433
- [Background] Park Y, Choi JE, Hwang HS. Protein supplementation improves muscle mass and physical performance in undernourished prefrail and frail elderly subjects: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2018 Nov 1;108(5):1026-1033. doi: 10.1093/ajcn/nqy214. PMID 30475969
- [Derived] Buhl SF, Beck AM, Christensen B, Caserotti P. Effects of high-protein diet combined with exercise to counteract frailty in pre-frail and frail community-dwelling older adults: study protocol for a three-arm randomized controlled trial. Trials. 2020 Jul 11;21(1):637. doi: 10.1186/s13063-020-04572-z. PMID 32653012